CLINICAL TRIAL: NCT01014871
Title: Intra-individual Comparison of the Efficacy of Two Botulinum Toxins Type A on Moderate to Severe Forehead Wrinkles After One Injection
Brief Title: Comparison of Two Botulinum Toxins Type A on Forehead Wrinkles
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.29081
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2012-04

CONDITIONS: Wrinkles
Keywords: Forehead Wrinkles Toxin
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- intra-individual comparison (Other)
  Interventions: Drug: Botulinum Toxin Type A - Azzalure; Drug: Botulinum Toxin Type A - Vistabel

INTERVENTIONS:
Drug: Botulinum Toxin Type A - Azzalure — One botulinum toxin type A will be injected in one side of the forehead and the other one will be injected in the other side of the forehead at Baseline. Allocation of each BoNT-A to each side of the forehead will be randomized.
Drug: Botulinum Toxin Type A - Vistabel — One botulinum toxin type A will be injected in one side of the forehead and the other one will be injected in the other side of the forehead at Baseline. Allocation of each BoNT-A to each side of the forehead will be randomized.

SUMMARY:
Single-centre, controlled, randomized, evaluator-blinded, bilateral (split-face) comparison study in subjects with moderate to severe forehead wrinkles.

One botulinum toxin type A will be injected in one side of the forehead and the other one will be injected in the other side of the forehead at baseline. Allocation of each BoNT-A to each side of the forehead will be randomized.

DETAILED DESCRIPTION:
There are two formulations of BoNT-A available: Botox®/Vistabel®, Allergan and Dysport®/Azzalure®, Ipsen - Galderma. These formulations behave distinctly in different ways electrophysiologically and clinically and results obtained with one formulation cannot be extrapolated to the other. There are only few clinical research directly comparing the two formulations in the treatment of forehead lines.

ELIGIBILITY:
Inclusion Criteria:

1. Female Subjects of any race, from 18 to 65 years old
2. Moderate to severe horizontal forehead wrinkles at maximum contraction (2-3 on the Forehead Wrinkles Severity Scale) on both sides of the forehead
3. Negative urine pregnancy test at the Baseline visit for Subjects of childbearing potential

Exclusion Criteria:

1. Subjects with a washout period for procedure(s)/treatment(s) on the forehead less than:

   * Retinoid, microdermabrasion, or prescription level glycolic acid treatments 2 weeks
   * Non-ablative light treatments (e.g. Intense Pulsed Light, light-emitting diodes) 1 month
   * Ablative skin resurfacing
   * Non-ablative dermal treatment for skin tightening (e.g. radio-frequency treatments) 6 months
   * Treatment with a BoNT-A 12 months
   * Soft tissue augmentation (e.g. biodegradable products as collagen or hyaluronic acid preparations) 24 months
2. Subjects who undergone a surgical facelift;
3. Permanent or semi-permanent dermal fillers in the forehead area;
4. Known allergy or hypersensitivity to any botulinum toxin or any component of BoNT-A (1) and/or BoNT-A (2) (see package inserts);
5. Concurrent use of treatments that affect neuromuscular transmission, such as curare-like depolarizing agents, lincosamides, polymyxins, anticholinesterases affecting the striated muscle and aminoglycoside antibiotics;
6. Pregnant women, nursing mothers, or women who are planning pregnancy during the study;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pr Rzany, MD, Principal Investigator — La Charité Hospital, Berlin, Germany
Locations (1):
- La Charité Hospital, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment process: patients from private practice - Recruitment period: First Patient In = 13 July 2009 Last Patient In = 09 November 2009 - Type of location: hospital
Groups:
- Vistabel/Azzalure: at Baseline:
  * 1 injection of 20 units of Azzalure (2 points of 10 units) in 1 side of the forehead
  * 1 injection of 8 Speywood units of Vistabel (2 points of 4 Speywood units) in the other side of the forehead
Period: Overall Study
Arm/Group | Vistabel/Azzalure
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vistabel/Azzalure
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Number; unit: participants]
  Germany | 30

OUTCOME MEASURES:

1. Primary Outcome: Severity of the Forehead Wrinkles by the Evaluator at Maximum Contraction and at Rest Using the Forehead Wrinkles Severity Scale (0 to 3) at Each Study Visit and for Each Side of the Forehead
Description: Bilateral comparison of forehead wrinkle severity score at rest and at maximum contraction measured by Forehead Wrinkles Severity Scale (0 to 3) at each study visit (Baseline, Days 1, 2, 3, 7, 10, 14, 30, Months 4 and 5)and for each side.
Time Frame: 5 months : Baseline, Days 1, 2, 3, 7, 10, 14, 30, Months 4 and 5
Population: Intention To Treat
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Azzalure: at Baseline:
  - 1 injection of 20 units of Azzalure (2 points of 10 units) in 1 side of the forehead
- Vistabel: at Baseline:
  - 1 injection of 8 Speywood units of Vistabel (2 points of 4 Speywood units) in the other side of the forehead
Arm/Group | Azzalure | Vistabel
Number analyzed (Participants) | 30 | 30
Scores on a scale
  Baseline at rest | 1.4 (0.5) | 1.4 (0.5)
  Day 1 at rest | 1.3 (0.5) | 1.3 (0.5)
  Day 2 at rest | 1.0 (0.6) | 1.0 (0.5)
  Day 3 at rest | 0.9 (0.6) | 0.8 (0.5)
  Day 7 at rest | 0.7 (0.7) | 0.7 (0.6)
  Day 10 at rest | 0.5 (0.6) | 0.5 (0.6)
  Day 14 at rest | 0.6 (0.6) | 0.5 (0.6)
  Day 30 at rest | 0.6 (0.6) | 0.6 (0.6)
  Month 4 at rest | 1.0 (0.5) | 1.0 (0.6)
  Month 5 at rest | 1.2 (0.6) | 1.3 (0.6)
  Baseline at maximum contraction | 2.1 (0.3) | 2.1 (0.3)
  Day 1 at maximum contraction | 1.8 (0.6) | 1.8 (0.6)
  Day 2 at maximum contraction | 1.6 (0.6) | 1.5 (0.6)
  Day 3 at maximum contraction | 1.2 (0.7) | 1.1 (0.6)
  Day 7 at maximum contraction | 0.7 (0.7) | 0.7 (0.7)
  Day 10 at maximum contraction | 0.6 (0.7) | 0.6 (0.6)
  Day 14 at maximum contraction | 0.5 (0.6) | 0.4 (0.5)
  Day 30 at maximum contraction | 0.5 (0.6) | 0.5 (0.5)
  Month 4 at maximum contraction | 1.5 (0.5) | 1.4 (0.6)
  Month 5 at maximum contraction | 1.8 (0.6) | 1.9 (0.5)

ADVERSE EVENTS:
Time Frame: 5 months
Description: All medical clinical events occurred after subject's consent signature and during the study, whether observed by the Evaluator/Injector or reported by the Subject and whether or not thought to be treatment-related were considered adverse events and collected.
Groups:
- Azzalure; Vistabel: intra-individual comparison
Arm/Group | Azzalure | Vistabel
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 15/30 | 18/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azzalure (N=30) | Vistabel (N=30)
DENTAL DISCOMFORT (Gastrointestinal disorders) | 2 (2) | 2 (2)
EYELID OEDEMA (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5)
EYELID PTOSIS (Eye disorders) | 2 (2) | 2 (2)
FACIAL PARESIS (Nervous system disorders) | 4 (4) | 4 (4)
HEADACHE (Nervous system disorders) | 4 (4) | 5 (5)
INJECTION SITE PARAESTHESIA (General disorders) | 1 (1) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 3 (3)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
SENSATION OF HEAVINESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
MIGRAINE (Nervous system disorders) | 2 (3) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreement in full force and effect for a period of 10 years.